CLINICAL TRIAL: NCT03001791
Title: Clinical and Histopathological Comparison of ER:YAG Laser, CO2 Laser and Scalpel Excision of Fibrous Hyperplasia on the Buccal Mucosa
Brief Title: Comparison of ER:YAG Laser, CO2 Laser and Scalpel Excision of Fibrous Hyperplasia on the Buccal Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 271-13
Record Dates: First submitted 2016-11-14; First posted 2016-12-23 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Fibrous Hyperplasia on Oral Mucosa
Keywords: CO2 laser; thermal damage zone; Er:YAG laser
MeSH Terms: interventions — Lasers, Solid-State; Lasers, Gas

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Er:YAG laser (Experimental): Excisional biopsy of fibrous hyperplasia with Er:YAG laser (Lite TouchTM, Synergon Dental Lasers, Light instruments Ltd., Yokneam Elite, Israel), λ = 2940nnm. Soft tissue biopsy mode with water cooling, frequency 35 Hz, pulse duration 250-390 µsec, pulse energy of 200 mJ, power 7 Watt . Cylindrical sapphire tip, 400 µm in diameter, without contact to the tissue.
  Interventions: Procedure: Excisional biopsy with Er:YAG laser
- CO2 laser (Experimental): Excisional biopsy of fibrous hyperplasia with CO2 laser (Spectra DENTA Surgical Carbon Dioxide Laser, MAX Engineering Ltd., Gyeonggi-Do, Korea), λ = 10'600nnm. cf mode (frequency 140 Hz, pulse duration 400 µsec, pulse energy 33 mJ,a power 4.62 watts). Laser beam with a spot size of 0.2 mm, non-contact mode.
  Interventions: Procedure: Excisional biopsy with CO2 laser
- Scalpel (Experimental): Excisional biopsy of fibrous hyperplasia with scalpel (blade 15C). Polyamide sutures (Seralon 5-DS15, Serag Wiessner KG, Naila, Germany).
  Interventions: Procedure: Excisional biopsy with scalpel

INTERVENTIONS:
Procedure: Excisional biopsy with Er:YAG laser — Excisional biopsy of fibrous hyperplasia in the buccal mucosa in local anesthesia with Er:YAG laser (Lite TouchTM, Synergon Dental Lasers, Light instruments Ltd., Yokneam Elite, Israel), λ = 2940nnm. Soft tissue biopsy mode with water cooling, frequency 35 Hz, pulse duration 250-390 µsec, pulse energy of 200 mJ, power 7 Watt . Cylindrical sapphire tip, 400 µm in diameter, without contact to the tissue.
  Arms: Er:YAG laser
Procedure: Excisional biopsy with CO2 laser — Excisional biopsy of fibrous hyperplasia in the buccal mucosa in local anesthesia with CO2 laser (Spectra DENTA Surgical Carbon Dioxide Laser, MAX Engineering Ltd., Gyeonggi-Do, Korea), λ = 10'600nnm. cf mode (frequency 140 Hz, pulse duration 400 µsec, pulse energy 33 mJ,a power 4.62 watts). Laser beam with a spot size of 0.2 mm, non-contact mode.
  Arms: CO2 laser
Procedure: Excisional biopsy with scalpel — Excisional biopsy of fibrous hyperplasia in the buccal mucosa in local anesthesia with scalpel (blade 15C). Polyamide sutures (Seralon 5-DS15, Serag Wiessner KG, Naila, Germany).
  Arms: Scalpel

SUMMARY:
The aim of the RCT is to analyse clinical and histopathological particularities for excisional biopsies of fibrous hyperplasia in the buccal mucosa performed with Er:YAG laser, CO2 laser and scalpel. The primary outcome parameter is to evaluate the thermal damage zone on the excised specimens. Secondary parameters are time of surgery, intraoperative bleeding, the need for additional electrocoagulation or sutures and patient's postsurgical perception of pain, other postsurgical effects and use of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Clinical tentative diagnosis of fibrous hyperplasia in the buccal mucosa
* Fibrous hyperplasia dimensions 0.5 to 2 cm
* Patient understands and reads the German language
* Written informed consent

Exclusion Criteria:

* Untreated diabetes Typ II
* Severe infectious disease (HIV, hepatitis)
* Severe psychiatric disease
* Immunosuppressive therapy
* Anticoagulation
* Pregnancy; a pregnancy test (Clearblue®) is performed in women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2017-07-04 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Histopathological thermal damage zone | Three months
  Biopsy specimens fixed in a 4% neutral-buffered formalin solution, embedded in paraffin, sectioned in slices of 5 μm, and stained with hematoxylin-eosin.
  Measurements of the thermal damage zone (in μm) on histopathological specimens by pathologist, blinded to the surgical method used. Measurements of the maximal and the minimal thermal damage zone on a representative section on both lateral edges of the fibrous hyperplasia.

SECONDARY OUTCOMES:
Postoperative Pain | Two weeks
  Registration of pain on VAS scale (ranging 0-100) during 14 days. The first VAS value was filled in before surgery, the second value in the evening after surgery and then on each of the following days on a study form handed out to patient.
  Intake of Analgesic (type, dose) are also filled in by patient on the study form i a specific section.
Number of patients with other postoperative effects | Two weeks
  Number of patients with other postoperative events (e.g. swelling, bleeding) on the same study form
Time of surgery | 15 minutes
  Registration of time of intervention with a stopwatch. It starts when the laser beam is first applied and ends when the wound paste had been applied.
Bleeding during surgery | 15 minutes
  Registration of bleeding events (yes/no) and method to stop the bleeding during surgery (electrocautery, sutures)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie GA Suter, Dr med dent, Principal Investigator — Department of Oral Surgery and Stomatology, Dental School, University of Bern
Locations (1):
- Department of oral Surgery and Stomatology, Dental school, University Bern, Bern, Switzerland

REFERENCES:
- [Derived] Suter VGA, Altermatt HJ, Bornstein MM. A randomized controlled trial comparing surgical excisional biopsies using CO2 laser, Er:YAG laser and scalpel. Int J Oral Maxillofac Surg. 2020 Jan;49(1):99-106. doi: 10.1016/j.ijom.2019.05.012. Epub 2019 Jun 21. PMID 31230766